CLINICAL TRIAL: NCT00356395
Title: Cardiovascular and Metabolic Effects of Combination Therapy With Ramipril and Candesartan In Hypertensive Patients
Brief Title: Safety and Effects of Ramipril Combined With Candesartan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-008
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2006-07-26 (Estimated); Status verified 2006-03

CONDITIONS: Hypertension
Keywords: endothelial function, insulin resistance, adipocytokines
MeSH Terms: conditions — Hypertension; Insulin Resistance | interventions — Ramipril; candesartan

INTERVENTIONS:
Drug: ramipril, candesartan

SUMMARY:
we hypothesized that combination therapy has additive beneficial effects to improve endothelial dysfunction and adipocytokine profiles in patients with hypertension.

DETAILED DESCRIPTION:
Forty patients will be given ramipril 10 mg and placebo, ramipril 10 mg and candesartan 16 mg, or candesartan 16 mg and placebo daily in a randomized, double-blind, placebo-controlled cross-over trial with three treatment arms and two washout periods (each 2 months).

ELIGIBILITY:
Inclusion Criteria:

* patients with mild to moderate hypertension

Exclusion Criteria:

* We will exclude patients with severe hypertension, unstable angina, acute myocardial infarction, or renal insufficiency.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-08; Study Completion 2006-03

PRIMARY OUTCOMES:
comparison of endothelium-dependent dilation among the 3 treatment schemes

CONTACTS AND LOCATIONS:
Overall Officials: Kwang K Koh, MD, Principal Investigator — Cardiology, Gil Heart Center, Gachon Medical School